CLINICAL TRIAL: NCT06029101
Title: Modalities of Surgical Treatment of Chiari Malformation Disease : Clinical Study and Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hamdy Hussein, demonistrator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chiari I surgical treatment
Record Dates: First submitted 2023-08-25; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Chiari Malformation, Type 1
MeSH Terms: conditions — Arnold-Chiari Malformation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chiari I malformation patients undergoing craniectomy (Experimental): modalities and outcomes of surgical treatment of chiari I malformation patients
  Interventions: Procedure: posterior fossa craniectomy with or without duraplasty

INTERVENTIONS:
Procedure: posterior fossa craniectomy with or without duraplasty — craniectomy of occipital bone and duroplasty with graft to expand the shallow posterior fossa and reposition the cerebellar tonsils.

SUMMARY:
Evaluation of postoperative outcomes of Chiari type I Malformation Patients at Department of Neurosurgery Assiut University Hospital .

DETAILED DESCRIPTION:
Chiari malformation is a group of craniocervical malformations involving the brain stem, cerebellum, upper spinal cord, and surrounding bony structure, encompassing a series of hindbrain herniation symptoms. The Austrian pathologist Hans Chiari ﬁrst described the malformation in 1891 and such abnormality is frequently identiﬁed in both young adult and pediatric patients.

There are four main types of chiari malformations with other subtypes. Chiari I malformation (CIM), in which the caudal poles of the cerebellar tonsils extend into the upper cervical spinal canal, is a common clinical type. Common clinical symptoms, including headache, altered sensation, weakness, dysphagia, sleep apnea.

Between 70% and 80% of patients with CIM have accompanying syringomyelia. Surgical treatment is widely accepted and is the only treatment chosen for symptomatic patients with Chiari malformations.

The aim of this study is to elucidate the most favorable procedures for CIM in terms of radiological and clinical outcomes.

Independent and dependent variables will be identiﬁed for analysis. The independent variables will include patient diagnosis, surgical techniques, patient age, patient chronic diseases and identified dependent variables including improvement of symptoms and signs, rates of intraoperative and postoperative adverse events, and perioperative mortality.

Different surgical modalities will be applied ,examples include bony decompression with or without duraplasty with the possibility of cerebellar tonsils resection (RT) .

Common complications include meningitis, CSF leak, pseudomeningocele, hydrocephalus, respiratory failure, hemorrhage, craniocervical instability, and/or death.

The outcome will be measured by reduction / increase of symptoms and signs using the Chicago Chiari outcome scale (CCOS).

ELIGIBILITY:
Inclusion Criteria:

* Chiari I Malformation patients who suffer from clinical symptoms and radiological manifestations.
* Patients fit for surgery

Exclusion Criteria:

* Other types of Chiari malformations
* Patients with multilevel cervical disc herniation .
* Patients with segmental instability .
* Patients unfit for surgery

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative outcomes of Chiari Malformation Patients at Department of Neurosurgery Assiut University Hospital . | 4 weeks postoperative
  using chicago chiari outcome score The Chicago Chiari Outcome Scale (CCOS) uses 4 postoperative outcome categories (pain, nonpain symptoms, functionality, and complications) graded 1 to 4 for a total possible score of 16 , when the score is higher ,it means better outcome. pain for example will be measured by Visual Analog Score for pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Taghian, professor, Study Chair — Assiut University; Ahmed Abdallah, Ass. prof, Study Director — Assiut University; Ismail Taha, lecturer, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Shamji MF, Ventureyra EC, Baronia B, Nzau M, Vassilyadi M. Classification of symptomatic Chiari I malformation to guide surgical strategy. Can J Neurol Sci. 2010 Jul;37(4):482-7. doi: 10.1017/s0317167100010507. PMID 20724256
- [Background] 2. Meadows J, Guarnieri M, Miller K, Haroun R, Kraut M, Carson BS. Type I Chiari malformation: a review of the literature. Neurosurg Q. 2001;11: 220-229.
- [Background] Hankinson T, Tubbs RS, Wellons JC. Duraplasty or not? An evidence-based review of the pediatric Chiari I malformation. Childs Nerv Syst. 2011 Jan;27(1):35-40. doi: 10.1007/s00381-010-1295-7. Epub 2010 Oct 2. PMID 20890606
- [Background] Dones J, De Jesus O, Colen CB, Toledo MM, Delgado M. Clinical outcomes in patients with Chiari I malformation: a review of 27 cases. Surg Neurol. 2003 Aug;60(2):142-7; discussion 147-8. doi: 10.1016/s0090-3019(03)00131-9. PMID 12900124